CLINICAL TRIAL: NCT05743257
Title: The UrbASanté Study
Brief Title: How Urban Interventions in Lower Socioeconomic Areas Influence Health Behaviors (UrbASanté Study)
Status: Recruiting | Type: Observational
Sponsor: Paris 12 Val de Marne University (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); University Gustave Eiffel (Other); National Research Agency, France (Other)
Responsible Party: Principal Investigator, Hélène Charreire, Assistant Professeur, Paris 12 Val de Marne University
Other Study IDs: University Paris Est Creteil
Record Dates: First submitted 2023-02-09; First posted 2023-02-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Health-Related Behavior
MeSH Terms: conditions — Health Behavior | interventions — Surveys and Questionnaires; Interviews as Topic; Air; Noise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental group: Volunteers living in a deprived neighborhood with urban transformations in Paris (France)
  Interventions: Behavioral: Questionnaire; Behavioral: Food diary supply; Behavioral: Interviews (semi-structured); Behavioral: air and noise
- Control group: Volunteers living in a deprived neighborhood without urban transformations in Paris (France).
  Interventions: Behavioral: Questionnaire; Behavioral: Food diary supply; Behavioral: Interviews (semi-structured); Behavioral: air and noise

INTERVENTIONS:
Behavioral: Questionnaire — Each participant completes a questionnaire (online or paper version) about socio-demographic characteristics, health outcomes (general health, respiratory health, and weight status), physical activity and sedentary behaviors, perception of neighborhood characteristics, air quality, and noise exposure.
Behavioral: Food diary supply — Sample of participant was issued with a food supply diary to record details of their household food supply and related trips over 1-mo period. Household food supply included food purchases, food gift/donation, and potential crops. For each food purchase, participants provided details of date, place of purchase and foods purchased (name, quantity and expense incurred). When till receipts were available in grocery stores or supermarkets, participants were asked to collect them in an envelope placed at the end of the food supply diary.
Behavioral: Interviews (semi-structured) — Sample of participants was interviewed about their food provisioning practice and living conditions.
Behavioral: air and noise — Sample of participant were instructed to wear air and noise sensors to record their daily environmental exposure for 7 consecutive days, except for sleeping, bathing and performing activities in the water. Particulate matter concentrations, the temperature, and the relative humidity were measured - the nitrogen dioxide (NO2) and ozone (O3) concentrations were determined with data loggers that integrate reliable electrochemical gas sensors. Noise levels was measured using noise dosimeters. Sensors were accompanied by an activity logbook in which participants were required to daily record time when awake and sleeping, and, if any, time and duration of workout or device removal

SUMMARY:
The UrbASanté study is a quasi-experimental research that aimed at assessing the impact of urban transformations (a natural experiment) in the health related behaviors, environmental exposure and perceived- health.

DETAILED DESCRIPTION:
The UrbASAnté study is an interdisciplinary project evaluating the relationships between urban transformations (urban regeneration programs) and health related behaviors, environmental exposure (air pollution, noise) and health (perceived) in a deprived neighborhood in Paris (France).

UrbASanté consists of quasi-experimental research (before/after protocol design) and includes an "exposed" group of inhabitants living in a neighborhood with urban transformation (intervention) and an "unexposed group" comprising inhabitants from neighborhood not undergoing urban changes (control).

Participants will be surveyed at enrollment and 24 months later.

ELIGIBILITY:
Inclusion Criteria:

* Living in areas with urban intervention in Porte de la Chapelle, Paris (for experimental group)
* Living in areas without direct urban interventions close to Porte de la Chapelle, Paris (for control group)
* Age above 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Porte de la Chapelle (Paris, France)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in the mean adequacy ratio (MAR) | at baseline and 24 month later
  Measure of individuals nutrient adequacy based on reported food intakes
Change in the mean excess ratio (MER) | at baseline and 24 month later
  Measure of excessive nutrient consumption, based on reported food intakes
Change in physical activity behaviors | at baseline and 24 month later
  Assessed by questions from the Sedentary, Transportation, and Activity Questionnaire (STAQ) with added questions about perception of active modes (walking and cycling). Using indicators of time spent in different transport modes (car or motorized vehicle, public transport, walking, cycling, other active transport) assessing the past-week frequency and duration of transport.
Change in sedentary behaviors | at baseline and 24 month later
  Assessed by questions from the Sedentary, Transportation, and Activity Questionnaire (STAQ) using indicator of past week sitting time spent during transport, leisure and work/study.
Change in perceived health | at baseline and 24 month later
  Assessed by the question "How is your health in general? Is it…" (very good/good/fair/bad/very bad) as a standard and cost-effective measure in health surveys.

SECONDARY OUTCOMES:
Age (in year) of each member of the household | at baseline
  Participants were asked to report the age of each member of the household.
Gender of adult members of the household | at baseline
  Participants were asked to report the gender of each adult of the household
Household income | at baseline
  Participants indicated their net income bracket of the household (by month)
Education level of each adult of the household | at baseline
  Participants were asked to report the highest education level achieved by each adult of the household (no degree, primary school, secondary school degree, bachelor degree, tertiary degree).
Living duration (in month/year) in the residential neighborhood | at baseline
  Participants were asked to indicate how long they had lived in the study area
Marital status | at baseline
  Participants were asked to report their marital status

CONTACTS AND LOCATIONS:
Overall Officials: Helene Charreire, Principal Investigator — Paris 12 Val de Marne University; Benoit Conti, Principal Investigator — University Gustave Eiffel
Locations (1):
- Université Paris Est Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Charreire H, Conti B, Bauchard L, Cisse NA, Perignon M, Rollet P, Perrin C, Blanchard S, Roda C, Feuillet T, Madelin M, Dupuis V, Evrard AS, Hellequin AP, Coll I, Larrue C, Baudet-Michel S, Vernouillet G, Ntsame-Abegue F, Fabre I, Mejean C, Oppert JM; UrbASante Study Group. A natural experiment to assess how urban interventions in lower socioeconomic areas influence health behaviors: the UrbASante study. BMC Public Health. 2023 Mar 15;23(1):498. doi: 10.1186/s12889-023-15388-2. PMID 36922807